CLINICAL TRIAL: NCT03983226
Title: A Phase II, Randomized Study of Cytoreductive Surgery Combined With Niraparib Maintenance in Platinum-sensitive, Secondary Recurrent Ovarian Cancer
Brief Title: Surgery and Niraparib in Secondary Recurrent Ovarian Cancer (SOC-3 Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Fudan University (Other); Shanghai Jiao Tong University School of Medicine (Other); Zhejiang Cancer Hospital (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGOG OV5; SGOG OV-05 (Other: Shanghai Gynecologic Oncology Group)
Record Dates: First submitted 2019-06-05; First posted 2019-06-12 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer Recurrent; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: reurrent Ovarian Cancer; Secondary Cytoreductive Surgery; Chemotherapy; Niraparib maintenance
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Surgical Procedures, Operative; Carboplatin; taxane; niraparib; Maintenance

STUDY DESIGN:
Intervention Model Description: randomized umbrella clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental): Intervention:
  Procedure: Maximum effort cytoreductive surgery combined with Niraparib maintenance Drug: Platinum-based chemotherapy and Niraparib
  Interventions: Procedure: Surgery; Drug: carboplatin/taxane, carboplatin/gemcitabine, cisplatin/gemcitabine, liposome doxorubicin/carboplatin...; Drug: Niraparib
- No surgery (Active Comparator): Intervention: Drug: Platinum-based chemotherapy and Niraparib
  Interventions: Drug: carboplatin/taxane, carboplatin/gemcitabine, cisplatin/gemcitabine, liposome doxorubicin/carboplatin...; Drug: Niraparib

INTERVENTIONS:
Procedure: Surgery — Tumor debulking surgery (surgery in recurrent ovarian disease)
  Other Names: secondary cytoreduction
  Arms: Surgery
Drug: carboplatin/taxane, carboplatin/gemcitabine, cisplatin/gemcitabine, liposome doxorubicin/carboplatin... — Salvage chemotherapy
  Other Names: third-line therapy
Drug: Niraparib — Niraparib maintenance therapy
  Other Names: maintenance therapy

SUMMARY:
This is a Phase II, open-label, multicenter, randomized umbrella study to evaluate the efficacy of cytoreductive surgery and Niraparib maintenance in participants with platinum-sensitive secondary recurrent ovarian cancer. Cohort 1 will focus on participants without prior use of PARP inhibitor, and without prior secondary cytoreduction (SCR) when first recurrence. Cohort 2 will focus on participants with prior use of PARP inhibitor, but without prior SCR when first recurrence. Cohort 3 will focus on participants with SCR when first recurrence, but without prior use of PARP inhibitor.

DETAILED DESCRIPTION:
This exploratory trial is to compare the efficacy of secondary cytoreductive surgery followed by chemotherapy and Niraparib maintenance, versus chemotherapy alone followed by Niraparib maintenance in patients with platinum-sensitive secondary recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years to ≤ 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients with platinum-sensitive, secondary relapsed epithelial ovarian, primary peritoneal, or fallopian tube cancer.
* Front-line or second-line treatment may have included maintenance therapy (i.e. bevacizumab, PARP inhibitor)

  * Cohort 1 and Cohort 3: No prior use of PARP inhibitor.
  * Cohort 2: Prior use of PARP inhibitor.
  * Cohort 3: No prior use of PARP inhibitor.
* Secondary cytoreductive surgery (SCR) when first recurrence

  * Cohort 1 and Cohort 2: Never received SCR
  * Cohort 2: Never received SCR
  * Cohort 3: Received SCR
* Assessed by the experienced surgeons, complete resection of all recurrent disease is possible. Single or localized lesions identified by CT, or MRI, or positron emission tomography/computed tomography (PET/CT). PI and Co-PI reach consensus if extensive lesions or carcinomatosis.
* It can be included if single lesion outside the peritoneal cavity can be resected.
* No more than 3 disease lesions by central-reviewed PET/CT imaging if the participated center has never participated in any surgical trials on ovarian cancer before.
* Patients who have given their signed and written informed consent and their consent.

Exclusion Criteria:

* Patients with borderline tumors as well as non-epithelial tumors.
* Patients for interval-debulking, or for second- or third-look surgery, or palliative surgery planned.
* Impossible to assess the resectability. Radiological signs suggesting complete resection is impossible.
* Patients who have received more than two previous regimen of chemotherapy (maintenance is not considered a third regimen).
* Third relapse or more.
* Patients with second or other malignancies who have been treated by surgery, if the treatment might interfere with the treatment of relapsed ovarian cancer or if major impact on prognosis is expected.
* Progression during chemotherapy or recurrence within 6 months after second-line platinum-based therapy
* Any contradiction not allowing surgery and/or chemotherapy and/or or Niraparib
* Accompanied by hypoxia serious chronic obstructive pulmonary disease
* Uncontrolled hypertension, cerebrovascular accident/ Stroke, myocardial infarct, unstable angina, untreated thrombosis, chronic congestive heart failure, or serious arrhythmia in need of medicine.
* Severe hepatitis, history of liver disease, nephrotic syndrome, renal insufficiency
* Active ulcer history, abdominal wall fistula, perforation of gastrointestinal tract, or Intra-abdominal abscess, or simultaneously apply treatment/prevent ulcers therapy.
* Uncontrolled diabetes
* Uncontrolled epilepsy need long-term antiepileptic treatment.
* Any medication induced considerable risk of surgery, e.g. estimated bleeding due to oral anticoagulating agents.
* ≥3 grade anemia, neutropenia or thrombocytopenia due to chemotherapy, and lasted for more than 4 weeks
* Patients with a known hypersensitivity to Niraparib or any of the excipients of the product.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
12-month disease non-progression rate | up to 12 months after last patient randomized
  12-month non-progression rate

SECONDARY OUTCOMES:
Progression-free survival | Up to 24 months after last patient randomized
  from date of randomization until the date of 3rd relapse/progression or death (whatever occurs first)
Treatment free survival | Up to 24 months after last patient randomized
  It is the area between Kaplan-Meier curves for two time-to-event end points: 1) time to protocol chemotherapy cessation and 2) time to first subsequent anticancer therapy initiation or death, whichever occurred first.
Overall survival | Approximately up to 24 months after last patient randomized
  from date of randomization until the date of death from any cause
30-day post-operative complications | From the operation until after 30 days
  surgical complications grading criteria will be adopted for evaluating the perioperative complications
Quality of life assessment | baseline; 6 and 12 months after randomization
  the European Organization for Research and Treatment (EORTC) core quality of life questionnaire (QLQ-C30, version 3.0) The total score (range from 0 to 1,000)

CONTACTS AND LOCATIONS:
Overall Officials: Tingyan Shi, M.D., Ph.D., Principal Investigator — Shanghai Gynecologic Oncology Group; Rongyu Zang, M.D., Ph.D., Study Chair — Shanghai Gynecologic Oncology Group
Locations (5):
- China (5):
  - Fudan University Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Fudan University, Shanghai
  - Shanghai Jiao Tong University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi T, Yin S, Zhu J, Zhang P, Liu J, Zhu Y, Wu S, Chen X, Wang X, Teng Y, Zhu T, Yu A, Zhang Y, Feng Y, Huang H, Bao W, Li Y, Jiang W, Zhang P, Li J, Ai Z, Zhang W, Jia H, Zhang Y, Jiang R, Zhang J, Gao W, Luan Y, Zang R. A phase II trial of cytoreductive surgery combined with niraparib maintenance in platinum-sensitive, secondary recurrent ovarian cancer: SGOG SOC-3 study. J Gynecol Oncol. 2020 May;31(3):e61. doi: 10.3802/jgo.2020.31.e61. PMID 32319233
- See also: Shanghai Gynecologic Oncology Group — http://www.ShanghaiGOG.org